CLINICAL TRIAL: NCT00960778
Title: Gender Differences in Response to Nicotine Replacement Therapy and De-Nicotinized Cigarettes
Acronym: BIRCWH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR#18333
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Nicotine Dependence
Keywords: gender; nicotine dependence; nicotine replacement therapy; extinction; denicotinized cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Coitus | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Women- denicotinized cigarette (Experimental): Treatment-seeking nicotine-dependent women will participate in functional magnetic resonance imaging (fMRI) with the presentation of smoking-related cues after four days of denicotinized cigarette (less than 0.5 gram nicotine) use.
  Interventions: Other: denicotinized cigarettes (Quest 3 cigarettes)
- Men- denicotinized cigarette (Experimental): Treatment-seeking nicotine-dependent men will participate in functional magnetic resonance imaging (fMRI) with the presentation of smoking-related cues after four days of denicotinized cigarette (less than 0.5 gram nicotine) use.
  Interventions: Other: denicotinized cigarettes (Quest 3 cigarettes)
- Women -nicotine patch (Experimental): Treatment-seeking nicotine-dependent women will participate in functional magnetic resonance imaging (fMRI) with the presentation of smoking-related cues under after receiving three days of a 21 mg nicotine patch.
  Interventions: Drug: nicotine patch (Nicoderm Committed Quitter (CQ), Habitrol)
- Men- nicotine patch (Experimental): Treatment-seeking nicotine-dependent men will participate in functional magnetic resonance imaging (fMRI) with the presentation of smoking-related cues under after receiving three days of a 21 mg nicotine patch.
  Interventions: Drug: nicotine patch (Nicoderm Committed Quitter (CQ), Habitrol)

INTERVENTIONS:
Drug: nicotine patch (Nicoderm Committed Quitter (CQ), Habitrol) — Nicotine patch 21 mg every 24 hours will be utilized for the three days after the first scanning session.
  Other Names: Nicoderm Committed Quitter (CQ); Habitrol; nicotine transdermal system; NRT
  Arms: Men- nicotine patch; Women -nicotine patch
Other: denicotinized cigarettes (Quest 3 cigarettes) — Cigarettes that contain trace levels of nicotine (less than .05 mg per cigarette) will be utilized ad lib in the study for 4 days after the nicotine patch.
  Other Names: Quest 3 cigarettes
  Arms: Men- denicotinized cigarette; Women- denicotinized cigarette

SUMMARY:
This study will investigate the underlying neurobiology of differences between male and female smokers. Research suggests that women are less responsive to nicotine replacement therapy (NRT) than men and more responsive to the sensory and behavioral aspects of smoking. This study proposed that male smokers will have a greater response to NRT demonstrated by reduced withdrawal symptoms, craving, and less blood-oxygen-level dependent functional magnetic resonance imaging (BOLD FMRI) regional brain activation in response to nicotine-cues as compared to female smokers treated with NRT. Additionally, female smokers will have a greater response to denicotinized cigarettes with decreased withdrawal symptoms, craving, and less BOLD fMRI activation in response to nicotine-cues as compared to male smokers.

DETAILED DESCRIPTION:
Women smokers are less responsive to nicotine replacement therapy (NRT) and more responsive to environmental cues associated with smoking behavior. This pilot study is designed to increase understanding of the neural circuitry underlying these differences. In the proposed study, adult male and female (10 per group) treatment-seeking nicotine-dependent individuals will participate in functional magnetic resonance imaging (fMRI) with the presentation of smoking-related cues under three conditions during a seven day period: baseline, after NRT, and after denicotinized cigarette facilitated-extinction. After baseline scanning, subjects will receive three days of 21 mg nicotine patch. Scanning procedures will be repeated on day 3. Subjects will then receive denicotinized cigarettes for ad lib smoking on days three through seven. Subjects will be asked to remain abstinent throughout the study period and they will be assessed daily with self-report, Carbon Monoxide (CO) monitor and for nicotine withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 - 60.
2. Meet criteria for primary nicotine dependence, smoke at least 70% of days in the last 30 days prior to assessment.
3. Participants will have afternoon end-expired carbon monoxide levels of at least 15 p.p.m. to confirm smoke inhalation.
4. Moderate to high levels of nicotine dependence confirmed by Fagerstrom Test of Nicotine Dependence score.
5. General good health confirmed by history & physical, serum chemistries, complete blood count, urinalysis, and electrocardiogram.
6. Able to read and understand questionnaires and informed consent.
7. Right-handed.
8. Treatment seeking.
9. Demonstrate subjective response to cues in a laboratory cue reactivity session.
10. Able to maintain abstinence from nicotine during the study period.
11. Participants must have a negative rapid-screening Urine Drug Screen (UDS) and pregnancy test prior to both imaging sessions and placement of the patch.
12. Female participants will use a reliable method of birth control throughout the study.

Exclusion Criteria:

1. Currently meets Diagnostic and Statistical Manual (DSM)-IV criteria for any other psychoactive substance dependence disorder except nicotine dependence.
2. Any psychoactive substance abuse within the last 30 days as evidenced by subject report or urine drug screen.
3. Use of other tobacco products.
4. Current use of nicotine replacement therapy or other smoking cessation treatment.
5. Meets DSM-IV criteria for current axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post-traumatic stress syndrome, bipolar affective disorder, schizophrenia, or any other psychotic disorder or organic mental disorder. The rationale for excluding them is that symptoms from these disorders may affect dependent variables and complicate interpretation of the data.
6. Current suicidal ideation with plan or homicidal ideation.
7. Need for maintenance or acute treatment with any psychoactive medication including antiseizure medications.
8. Clinically significant medical problems such as cardiovascular, renal, GI, or endocrine problem that would impair participation or limit ability to participate in scan.
9. Sexually active females of child-bearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
10. Has current charges pending for a violent crime (not including Drive Under Influence (DUI) related offenses).
11. Persons with ferrous metal implants or pacemaker since fMRI will be used.
12. Persons who live with another smoker who is unwilling or unable to refrain from smoking in the home or presence of the participant.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hartwell, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine- Dependent Women: Over a period of one week, nicotine-dependent women completed 3 scans while being shown smoking related cues. Participants completed a baseline scan, a scan following 3 days of Nicotine Replacement Therapy (21 mg nicotine patch), and one following 4 days of denicotinized cigarette use.
- Nicotine- Dependent Men: Over a period of one week, nicotine-dependent men completed 3 scans while being shown smoking related cues. Participants completed a baseline scan, a scan following 3 days of Nicotine Replacement Therapy (21 mg nicotine patch), and one following 4 days of denicotinized cigarette use.
Period: Overall Study
Arm/Group | Nicotine- Dependent Women | Nicotine- Dependent Men
Started | 17 | 16
Completed | 8 | 13
Not Completed | 9 | 3

BASELINE CHARACTERISTICS:
Population: Participants were enrolled in the study and underwent baseline scanning procedures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine- Dependent Women | Nicotine- Dependent Men | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 0 | 17
  Male | 0 | 16 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 1 | 6
  White | 10 | 14 | 24
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Post- Cue Exposure Craving Nicotine Patch
Description: Participants will complete cue exposure sessions after 3 days of nicotine patch use and rate craving on a 10 item self-report questionnaire. The Within Sessions Rating scale measures craving with 0 indicating Not at All and 10 indicating Extremely.
Time Frame: Day 3
Population: 12 women and 15 men completed the 3 days of Nictoine Replacement Therapy and completed the second scan.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine- Dependent Women | Nicotine- Dependent Men
Number analyzed (Participants) | 12 | 15
score on a scale | 25.58 (14.82) | 25.6 (12.6)

2. Primary Outcome: Post- Cue Exposure Craving Denicotinized Cigarettes
Description: Participants will complete cue exposure sessions after 4 days of denicotinized cigarette us and rate craving on a 10 item self-report questionnaire, the Questionnaire of Smoking Urges- Brief (QSU-B). Participants rate craving on a scale on a 1-7 point Likert scale where indicates Strongly Disagree and 7 indicates Strongly Agree. Higher scores indicate higher craving. Ratings from the 10 items are summed to attain the score reported here.
Time Frame: Day 7
Population: 8 women and 13 men complete the 4 days of denicotinized cigarette use and completed the third scan.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine- Dependent Women | Nicotine- Dependent Men
Number analyzed (Participants) | 8 | 13
score on a scale | 22.13 (14.38) | 17.85 (9.21)

ADVERSE EVENTS:
Arm/Group | Nicotine- Dependent Women | Nicotine- Dependent Men
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes